CLINICAL TRIAL: NCT00006377
Title: Phase II Study of Sequential Administration of Doxorubicin, Paclitaxel, and Carboplatin in Patients With Advanced and Recurrent Endometrial Cancer
Brief Title: Doxorubicin, Paclitaxel, and Carboplatin in Treating Patients With Primary Stage III, Stage IV, or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-073; CDR0000068251 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1860
Record Dates: First submitted 2000-10-04; First posted 2003-05-30 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Endometrial Cancer
Keywords: stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Doxorubicin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: doxorubicin hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining doxorubicin, paclitaxel, and carboplatin in treating patients who have primary stage III, stage IV, or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and duration of response in patients with primary stage III or IV or recurrent endometrial cancer treated with sequential doxorubicin, paclitaxel, and carboplatin.

OUTLINE: Patients receive sequential chemotherapy comprised of doxorubicin IV once every 2 weeks for 3 courses, followed by paclitaxel IV over 1 hour once weekly for 9 courses, and then carboplatin IV once every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 18-46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven primary stage III or IV or recurrent endometrial cancer
* Bidimensionally measurable disease by x-ray, CT scan, MRI scan, or physical exam

  * Sole site may be within a previously irradiated area if documented disease progression since prior radiotherapy

PATIENT CHARACTERISTICS:

Age:

* Adult

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin, SGOT, and alkaline phosphatase no greater than 1.5 times normal

Renal:

* Creatinine no greater than 1.8 mg/dL

Cardiovascular:

* Left ventricular ejection fraction at least 50%

Other:

* No active uncontrolled infection
* No greater than grade II neuropathy
* No other active malignancy
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior doxorubicin
* Greater than 6 months since prior paclitaxel, carboplatin, or other platinum compounds

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States